CLINICAL TRIAL: NCT04464785
Title: CentriMag Failure-to-Wean Post-Approval Study
Brief Title: CentriMag Failure-to-Wean Post Approval Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10336
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment: Subjects who receive the CentriMag Circulatory Support System
  Interventions: Device: CentriMag Circulatory Support System

INTERVENTIONS:
Device: CentriMag Circulatory Support System — The CentriMag Circulatory Suppose System is indicated for providing support for up to 30 days for one or both ventricles of the heart to treat post-cardiotomy patients who fail-to-wean from cardiopulmonary bypass, providing a bridge to decision when it is unclear whether the patient's heart will recover or whether the patient will need alternative, longer-term therapy.

SUMMARY:
The primary objective of this Post Approval Study is to report the proportion of patients surviving to 30 days post CentriMag support or to hospital discharge, whichever is longer. For subjects who do not recover and are bridged to a heart transplant or a long-term assist device, the primary endpoint is survival to induction of anesthesia for the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject >18 years of age
* Subject or legal representative has signed Informed Consent Form (ICF)
* Subject has CentriMag Circulatory Support System implanted due to Failure To Wean from Cardiopulmonary Bypass

Exclusion Criteria:

• Concomitant use of Extracorporeal Membrane Oxygenation (ECMO) during CentriMag Circulatory Support System implantation due to FTW from CPB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects who fail-to-wean from cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Survival to 30 days Post CentriMag support or to hospital discharge | 30 days
  The proportion of subjects who survive to 30 days post CentriMag support or to hospital discharge (whichever is longer).
Survival to induction of anesthesia for surgery for transplant or a long-term system | Approximately 30 days
  The proportion of subjects who do not recover and are bridged to a transplant or long-term system

CONTACTS AND LOCATIONS:
Overall Officials: Brian Crowe, Study Director — Abbott
Locations (8):
- United States (8):
  - Baptist Healt Medical Center, Little Rock, Arkansas
  - Emory University Hospital, Atlanta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No